CLINICAL TRIAL: NCT04445363
Title: A Phase I/II Study Of The Efficacy,Safety and Pharmacokinetics Of Jaktinib Hydrochloride Cream In Subjects With Mild To Moderate Alopecia Areata
Brief Title: A Study With Jaktinib Hydrochloride Cream Applied Topically to Subjects With Alopecia Areata
Acronym: AA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAKT001
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Alopecia Areata(AA)
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: In phase I of this study, Forty enrolled subjects were randomly assigned to four groups at 1:1:1:1. (1) concentration of 0.5%, twice daily (Bid) group; (2) concentration of 1.5%, bid group; (3) concentration of 2.5%, once daily(Qd) group; (4) concentration of 2.5%, bid group.Ten subjects in each group were randomly assigned to receive Jaktinib hydrochloride cream (8 cases) and placebo (2 cases) at 4:1, respectively,The duration of administration was 24 weeks.
  In phase II of this trial, 120 Enrolled subjects are randomly assigned to 3 groups (placebo bid group,concentration of 1.5% bid group and concentration of 2.5% bid group).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1,0.5% Bid (Experimental): Jaktinib hydrochloride cream 0.5% concentration, twice daily
  Interventions: Drug: Jaktinib hydrochloride cream
- Cohort 1,1.5% Bid (Experimental): Jaktinib hydrochloride cream 1.5% concentration, twice daily
  Interventions: Drug: Jaktinib hydrochloride cream
- Cohort 1,2.5% Qd (Experimental): Jaktinib hydrochloride cream 2.5% concentration, once daily
  Interventions: Drug: Jaktinib hydrochloride cream
- Cohort 1,2.5% Bid (Experimental): Jaktinib hydrochloride cream 2.5% concentration, twice daily
  Interventions: Drug: Jaktinib hydrochloride cream
- Dose extension: Placebo (Placebo Comparator): Placebo, twice daily
  Interventions: Drug: Placebo
- Dose extension: 1.5% Bid (Experimental): Jaktinib hydrochloride cream 1.5% concentration, twice daily
  Interventions: Drug: Jaktinib hydrochloride cream
- Dose extension: 2.5% Bid (Experimental): Jaktinib hydrochloride cream 2.5% concentration, twice daily
  Interventions: Drug: Jaktinib hydrochloride cream

INTERVENTIONS:
Drug: Jaktinib hydrochloride cream — Jaktinib hydrochloride cream/placebo applied topically in the morning and in the evening, administered continuously for 24 weeks
  Other Names: Jaktinib
  Arms: Cohort 1,0.5% Bid; Cohort 1,1.5% Bid; Cohort 1,2.5% Bid; Cohort 1,2.5% Qd; Dose extension: 1.5% Bid; Dose extension: 2.5% Bid
Drug: Placebo — Dose extension: Placebo
  Arms: Dose extension: Placebo

SUMMARY:
This study includes a dose escalation part(phase I) and a dose extension part(phase II).

DETAILED DESCRIPTION:
In phase I of this study, a multi-center, randomized, placebo parallel control design was adopted. Enrolled subjects were randomly assigned to the experimental group or the placebo group.A total of 40 subjects are expected to be enrolled in about 4 centers.

In phase II of this study, a multi-center, randomized, double-blind parallel, placebo-controlled design was adopted. Enrolled subjects were randomly assigned to the experimental group or the placebo group.About 120 subjects are expected to be enrolled in about 10 centers.

ELIGIBILITY:
Inclusion Criteria:

* 18 ~ 65 years old (including boundary value), regardless of gender;
* Diagnosis of Alopecia Areata;
* Hair loss accounts for 5% ~ 49% of the total scalp area;
* The duration of hair loss is at least 6 months, the longest is not more than 5 years;
* Patients can complete treatment for at least 6 months;
* About Fertility needs meet the following criteria: The results of serum pregnancy tests performed by fertile women during screening visits must be negative, and the results of human chorionic gonadotropin tests performed before the initiation of the study drug must be negative;Women who were fertile and men who had not received vasectomies were required to use effective contraception throughout the study period beginning with the informed consent and up to six months after the last administration;
* Subjects will voluntarily participate in the study after learning about the content and potential adverse drug reactions and must sign an IRC-approved informed consent prior to beginning any examination required by the study;
* Subject is willing and able to comply with scheduled visits, treatment plan, study drug administration, and other study procedures.

Exclusion Criteria:

* The following causes of hair loss should be excluded: hair loss caused by androgenic alopecia,syphilis, thyroid diseases, etc.
* Acute Diffuse and Total Alopecia of the Female Scalp;
* Prior history of serious chronic diseases, such as thyroid disease, liver disease, malnutrition, heart disease, nervous system disease, gastrointestinal dysfunction, tumor and mental illness, etc;
* Human immunodeficiency virus infection, hepatitis C virus infection, hepatitis B virus infection;
* Participated in a trial for a topical or oral JAK inhibitor;
* Allergic reactions to active ingredients or excipients are known or determined by the investigator;
* Receipt of treatment known to potentially affect the course of AA within last 3 month;
* In the opinion of the investigator , the subject is inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving 90% Improvement of Severity of Alopecia Tool (SALT90) | at week 24
  SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 90 response is a 90% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease.

SECONDARY OUTCOMES:
Change in Severity of Alopecia Tool (SALT) Score | at baseline, at week 12 and at week 24
  Severity of Alopecia Tool Score (SALT) calculation is based on a scoring system. The scalp is divided into the following 4 areas: 1) Vertex: 40% (0.4) of scalp surface area, 2) Right profile of scalp: 18% (0.18) of scalp surface area, 3) Left profile of scalp: 18% (0.18) of scalp surface area, and 4) Posterior aspect of scalp: 24% (0.24) of scalp surface area. The percentage of hair loss in any of these areas is the percentage hair loss multiplied by percent surface area of the scalp in that area. The SALT score is the sum of percentage of hair loss in all the above-mentioned areas, so a lower number indicates a better outcome. The reported SALT score range is from a minimum of 0 (no hair loss) to a maximum of 100 (100% hair loss).

CONTACTS AND LOCATIONS:
Overall Officials: qianjin lu, M.D., Study Chair — The Second Xiangya Hospital, Central South University
Locations (1):
- The Second Xaingya Hospital，central south university, Changsha, Hunan, China